CLINICAL TRIAL: NCT03128073
Title: A Feasibility Study of Peritoneal Ultrafiltration With a Wearable Device, CLS UF, That Adds a Glucose-salt Solution to the Intraperitoneal Fluid in the Device, in Order to Maintain a Stable Intraperitoneal Osmolarity and Thereby Enhance Ultrafiltration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Triomed AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Tmed-004 (Malmö)
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Ultrafiltration Failure
Keywords: Heart failure, Cardio-Renal Syndrome
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome | interventions — Ultrafiltration

STUDY DESIGN:
Intervention Model Description: Intervention study, pilot/ feasibility for proof of concept of peritoneal ultrafiltration with the Carry Life system ultrafiltration (CLS UF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): The intervention is with the Carry Life system ultrafiltration (CLS UF) device, which administers a Glucose-salt solution intermittently to a volume of the intraperitoneal fluid in the device.
  Interventions: Device: Carry life system, ultrafiltration (CLS UF)

INTERVENTIONS:
Device: Carry life system, ultrafiltration (CLS UF) — The addition of Glucose-salt intermittently to a volume of the intraperitoneal fluid in the device which is then returned to the subject.

SUMMARY:
The study is a proof-of-concept, a feasibility study of peritoneal ultrafiltration with a wearable device, Carry Life System Ultrafiltration (CLS UF) and will be performed on 4-6 stable peritoneal dialysis (PD) patients without clinical signs of dehydration. The study session starts with an initial fill of the abdomen, with a standard, glucose based PD solution. The CLS UF device is then connected to the patients existing, PD catheter. A Glucose-salt solution is added to 180 ml of the intraperitoneal fluid which is intermittently transferred from the peritoneal cavity through a closed system using the CLS UF cycler and then returned to the patient. The addition of the Glucose-salt solution maintains a stable intraperitoneal osmolarity and compensates for the glucose uptake and dilution which occurs in standard PD treatments.

DETAILED DESCRIPTION:
At visit 1: the fulfilment of the inclusion criteria. a medical assessment including vital signs, and a written informed consent are obtained. A peritoneal equilibrium test (PET) is performed at visit 2, which is a semi-quantitative assessment of peritoneal membrane transport function in patients on peritoneal dialysis. The PET test will determine if the subject has a low, medium or high transport capacity which in turn will dictate the Glucose-salt setting required in the CLS UF to achieve the desired ultrafiltration volume. The dosage of the Glucose-salt solution is based on an algorithm and according to the algorithm, the target osmolarity should be 340 mOsmol/L to obtain an ultrafiltration flow rate of approximately 150 ml/h.

The study session with the CLS UF will be performed both at visit 3 and 4. If the prescription of the glucose-salt solution has been changed between treatment sessions 1 and 2 there is an option of a 5th visit. The patient will perform the ordinary prescribed PD therapy until the evening before the study session day, according to the prescription of the investigator. The abdomen will be without PD solution during the night. On the morning of the study day an initial assessment of the patient will be performed before starting the study session and thereafter the abdomen will be filled with a fresh of PD solution, immediately followed by a complete drain.

The study session starts with a fill of the abdomen with 2000 ml of Physioneal 2.27%. The sodium concentration of the glucose-salt solution and the glucose dosage required to achieve the target osmolarity of 340 mOsm/L in the intraperitoneal fluid is set according to the Glucose dosage table (CIP, Table 3). The CLS UF device will then be connected to the catheter via the patient line and the device started. The study session is performed for 8 hours and Intermittent drains of 180 ml intraperitoneal fluid will be performed hourly to maintain a stable intraperitoneal volume of around 2 liters. A new cycle starts directly after each drain. The patient can at any time start an extra drain if he/she experience discomfort of increased volume in the abdomen. At the end of the session a complete drain of the peritoneal cavity will be performed and the volume measured. During the study session blood and dialysate samples will be taken according to the case report form (CRF). During the study session, the subjects will eat and drink as usual. All intakes and outputs of fluids will be measured. After the completed study sessions (visit 3 & 4), the Investigator will perform a clinical assessment of the patient and if satisfactory the patient will return home.

At visit 6, a follow up visit is performed in which the subject's vital signs are performed. Adverse events are assessed during study session between visit 3 and follow-up (visit 6). An evaluation of the treatment sessions by the subjects is also performed from visit 3 to visit 6.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, of more than 18 years of age.
* Prevalent PD patients without clinical signs of dehydration.
* Obtained written consent to participate in the study.

Exclusion Criteria:

* Active malignant disease.
* On-going infection.
* HIV and/or hepatitis positive.
* Pregnant, breastfeeding or women of childbearing potential without adequate contraceptive precautions.
* Diabetes type 1.
* Abdominal hernias.
* Conditions except the previous that the Investigator assesses as unsuitable for participation.
* Participation in other clinical trials, which can interfere with this study, within one month before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Osmolarity in the intraperitoneal fluid and Ultrafiltered volume during a study session. | Eight hour study session
  Ultrafiltration during the eight hour study session.
Ultrafiltered volume during a study session. | Eight hour study session
  To calculate the total ultrafiltration volume both the total fluid intake and the total output will be calculated during the study session. The fluid intake is recorded and subtracted from the total output which consists of: hourly drains, dialysate sample volumes, the total drain of the peritoneal cavity and the urinary output.

SECONDARY OUTCOMES:
Electrolyte gap, i.e. the difference between the electrolyte removal (Na+, K+, Ca++, Mg++) calculated theoretically for an isotonic ultrafiltration fluid and the amount actually removed. | During eight hour study session
  Measurement of electrolytes in serum and intraperitoneal fluid during the study session.
The patient will verbally evaluate the treatment with the CLS UF and give there subjective opinion of the wearable device. | During eight hour study sessions and in the follow-up visit
  The patient will verbally evaluate the treatment with the CLS UF (e.g. related to the intermittent transfer of intraperitoneal fluid in and out of the device). The patient give their subjective opinion of the wearable device (e.g. related to the weight, ease of movement, comfort etc.)
The incidence of treatment emergent adverse events or adverse device events occurring from the start of the first study session (Visit 3) until the last follow up visit will be evaluated and reported. | From the third study visit to the completion of the follow-up visit
  Electrolytes and glucose will be measured both in the blood and the intraperitoneal fluid during the study sessions. The incidence of treatment emergent adverse events or adverse device events occurring from the start of the first study session (Visit 3) until the last follow up visit will be evaluated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Cathrine Johansson, MD, PhD, Principal Investigator — Skånes University Hospital Malmö, Renal Unit, Inga-Marie Nilsson Gatan, 205 02 Malmö
Locations (1):
- Kidney Unit, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No